CLINICAL TRIAL: NCT00478400
Title: Awareness of Deficit After Combat-related Brain Injury
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: NEUC-029-06S; H-2006-0256 (Other Grant/Funding Number: University of Wisconsin, Madison)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Traumatic Brain Injury; Veterans
Keywords: Recovery; Magnetic resonance imaging; Awareness; Neurologic deficits
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Participants who have had a TBI: (recruited by invitation only)
  1. Must be between 1- and 6-years post-injury
  2. Closed head injury
  3. Evidence of loss of consciousness
  4. Must have an informant (friend, spouse, child etc.)
  5. Audit-C < 7, PCL < 65 and PHQ-9 < 15
- Participants with No history of TBI: (Recruited by invitation only)
  1. No history of TBI
  2. Must have an informant (friend, spouse, child etc.)
- Veterans with History of TBI: 1. Must be between 1- and 6-years post-injury
  2. Closed head injury
  3. Evidence of loss of consciousness
  4. Must have an informant (friend, spouse, child etc.)
  5. Audit-C < 7, PCL < 65 and PHQ-9 < 15
- US Veterans with No history of TBI: 1. No history of TBI
  2. Must have an informant (friend, spouse, child etc.)

SUMMARY:
This study will use MRI imaging, cognitive testing and outcome questionnaires to determine how the brain recovers and reorganizes after an injury.

DETAILED DESCRIPTION:
The extent of recovery from brain injury is often difficult to predict because of our limited understanding of how the brain changes as it heals. New brain imaging methods may help in this regard. One imaging technique called functional magnetic resonance imaging (fMRI) has made it possible to study the brain "at work"; that is, we can see regions of the brain that are active during particular tasks such as focusing attention, making decisions, or remembering words and pictures. Another MRI method called diffusion tensor imaging provides information on the pathways between brain regions that may be altered with brain injury.

The goals of this research are to 1) determine the brain regions involved in making accurate judgments about one's abilities and disabilities after a brain injury and whether damage to these brain areas affects outcome; and 2) examine how recovery of cognitive and physical abilities relates to changes in brain function over time. In order to accomplish the first goal we will recruit Veterans who have sustained a head injury and matched control subjects. For the second goal, we are asking patients and controls who have previously participated in brain injury research with our lab to come back for another visit at three years post-injury.

ELIGIBILITY:
Inclusion Criteria:

* History of traumatic brain injury at least 12 months prior to enrollment
* Control Group: No history of traumatic brain injury

Exclusion Criteria:

* Claustrophobia
* Metallic or electronic implants or devices that are not MRI-safe
* Foreign metal, such as shrapnel, in the body

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Veterans will be recruited through the Middleton VA Hospital in Madison, WI. Civilian participants will be recruited from a previous study led by Dr. Johnson.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Cognition change at study endpoint between TBI and controls | Greater than 3 years post-injury
Longitudinal change in white matter | 2 months, 1 year, and greater than 3 years post-injury
  Participants will include post-TBI in survivors the investigators have studied previously
Longitudinal change in whole brain morphology | 2 months, 1 year, and greater than 3 years post-injury
  Participants will include post-TBI in survivors the investigators have studied previously

CONTACTS AND LOCATIONS:
Overall Officials: Sterling C Johnson, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States